CLINICAL TRIAL: NCT06515262
Title: A Clinical Study to Evaluate the Safety and Efficacy of BCMA-GPRC5D CAR-T in Patients With Relapsed/Refractory Multiple Myeloma Who Received Three or More Lines of Therapy
Brief Title: Safety and Efficacy of Anti-BCMA-GPRC5D CAR-T Cells Therapy in the Treatment of r/r MM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China (Other)
Collaborators: Guangzhou Bio-gene Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BG-CT-23-015
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Relapsed/Refractory Multiple Myeloma
Keywords: BCMA-GPRC5D CAR-T
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-BCMA CAR-T (Experimental): BCMA-GPRC5D CAR-T is a novel CAR cell therapy for the treatment of relapsed/refractory multiple myeloma.
  Interventions: Biological: Anti-BCMA-GPRC5D CAR-T cells infusion

INTERVENTIONS:
Biological: Anti-BCMA-GPRC5D CAR-T cells infusion — Subiects who meet the enrollment conditions will receive intravenous infusion of anti-BCMA-GPRC5D CAR-T Cells after lymphodepleting therapy.

SUMMARY:
This is a single-center, open-label, single-arm study to evaluate the safety and efficacy of bispecific BCMA-GPRC5D CAR-T cells in patients with relapsed or refractory multiple myeloma who received three or more lines of therapy.

DETAILED DESCRIPTION:
This is a single-center, open-label, single-arm study to evaluate the safety and efficacy of bispecific BCMA-GPRC5D CAR-T cells in patients with relapsed or refractory multiple myeloma who received three or more lines of therapy.A leukapheresis procedure will be performed to manufacture Anti-BCMA-GPRC5D chimeric antigen receptor (CAR) modified T cells. Prior to Anti-BCMA-GPRC5D CAR-T cells infusion subjects will receive lymphodepleting therapy with fludarabine and cyclophosphamide. After infusion, the safety and efficacy of CAR-T therapy was evaluated by investigators.

ELIGIBILITY:
Inclusion Criteria:

1. The patient or his/her guardian understands and voluntarily signs the informed consent, and is expected to complete the follow-up examination and treatment of the study procedure;
2. Age 18-75 years old, gender unlimited;
3. Diagnosed as Multiple Myeloma (MM) according to the international standard for multiple myeloma (IMWG);
4. The presence of measurable disease at screening meets one of the following criteria:Serum M-protein ≥ 1.0 g/dL or Urine M-protein ≥ 200 mg/24h or diagnosed as Light-chain MM without measurable disease in serum and urine; Serum free light chain ≥ 10 mg/dL with an abnormal κ/λ ratio;
5. Patients must relapse or be refractory after three or more lines of therapy, which at least include: one Proteasome Inhibitor (PI), one Immunomodulatory Drug (IMiD), and one anti-CD38 monoclonal antibody;
6. diagnosed as relapsed/refractory disease or primary refractory disease;
7. The last treatment is ineffective, or the disease progresses within 60 days after the end of the last therapy;
8. The patient has recovered from the toxicity of the prior treatment, i.e., CTCAE toxicity grade < 2 (unless the abnormality is related to the tumor or is stable as judged by the investigator and has little impact on safety or efficacy);
9. ECOG score 1-2 points and the expected survival period ≥ 3 months;
10. Liver, kidney and cardiopulmonary functions meet the following requirements:

    1. Total bilirubin ≤ 1.5×ULN, alanine aminotransferase (ALT) ≤ 3 × ULN and aspartate aminotransferase (AST) ≤ 3 × ULN;
    2. Serum creatinine ≤ 1.5×ULN, or creatinine clearance ≥ 60 mL/min;
    3. Hemoglobin (Hb) ≥ 50 g/L without prior blood transfusion within 7 days;
    4. Baseline peripheral oxygen saturation > 92%;
    5. Corrected serum calcium ≤ 12.5 mg/dL (≤ 3.1 mmol/L) or free (ionized, ionic) calcium ≤ 6.5 mg/dL (≤ 1.6 mmol/L);
    6. Left ventricular ejection fraction (LVEF) > 45%, without confirmed pericardiac effusion and abnormal electrocardiography with clinical significance;
    7. Without clinically significant pleural effusion;
11. Venous access could be established; without contraindications of apheresis.

Exclusion Criteria:

1. Have been diagnosed with or treated for aggressive malignancies other than multiple myeloma;
2. Prior antitumor therapy (prior to blood collection for CAR-T preparation) : targeted therapy, epigenetic therapy, or investigational drug therapy within 14 days or at least 5 half-lives, whichever is shorter;
3. It is suspected that MM has involved the central nervous system or meninges and has been confirmed by MRI or CT, or there are other active central nervous system diseases;
4. Patients with Fahrenheit macroglobulinemia, POEMS syndrome, or primary AL, amyloidosis;
5. Subjects with positive HBsAg or HBcAb positive and peripheral blood HBV DNA titer is higher than the lower limit of detection of the research institution; HCV antibody positive; HIV antibody positive; CMV DNA titer is higher than the lower limit of detection of the research institution; EBV DNA titer is higher than the lower limit of detection of the research institution;
6. Patients have a severe allergic history;
7. Any unstable systemic disease: including but not limited to unstable angina, cerebrovascular accident or transient cerebral ischemia (within 6 months before screening), myocardial infarction (within 6 months before screening), congestive heart failure [New York Heart Association (NYHA) classification ≥ grade III];
8. Systemic diseases judged by researchers to be unstable: including but not limited to severe liver, kidney or metabolic diseases requiring drug treatment;
9. Patients with acute/chronic graft-versus-host disease (GVHD) or requiring immunosuppressive therapy for GVHD within 6 months prior to screening;
10. Active autoimmune or inflammatory diseases of the nervous system;
11. Patients develop oncology emergencies and need to be treated before screening or infusion;
12. Uncontrolled infections that need antibiotics treatment;
13. Exposure to hematopoietic growth factor of cells within 1-2 weeks before apheresis;
14. Exposure to Corticosteriods or immunosuppressive agents within 2 weeks before apheresis;
15. Patients receive a major surgical operation within 4 weeks before lymphodepletion or do not recover completely before the enrollment; or plan to receive a major surgical operation during the study period;
16. Live attenuated vaccine within 4 weeks before screening;
17. Persons with serious mental illness;
18. Alcoholics or persons with a history of drug abuse;
19. Pregnant or Lactating Women; Patients and his or her spouse have a fertility plan within two years after CAR-T cell infusion;
20. Any unsuitable to participate in this trial judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events(AE) after infusion | within 2 years after infusion
  The frequency, severity, and laboratory findings of all adverse events/serious adverse events are included.Cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome are graded by American Society for Transplantation and Cellular Therapy (ASTCT) criteria.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | within 2 years after infusion
  Overall Response Rate (ORR) is defined as the proportion of subjects achieving strict complete remission(sCR), complete response(CR), very good partial response(VGPR） and partial response(PR).
Concentration of CAR-T cells | Days 1,4, 7, 10, 14 ,21,28and months 2, 3, 6, 9, 12,18,24 after infusion
  Concentration of CAR-T cells measured by Flow cytometry after CAR-T infusion
Progression-free survival(PFS) | within 2 years after infusion
  Progression-free survival(PFS) refers to the time from cell reinfusion to the first assessment of tumor progression or death from any cause.
Overall survival(OS) | within 2 years after infusion
  Overall survival (OS) refers to the time from the time the patient received an infusion of CAR-T cells until death (from any cause).

CONTACTS AND LOCATIONS:
Overall Officials: Sanbin Wang, Principal Investigator — 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China
Locations (1):
- Sanbin Wang, Kunming, Kunming, Yunnan, China